CLINICAL TRIAL: NCT04574544
Title: Pilot Zinc Supplementation and Nutrition Education Among Children in the Rural Community, Cameroon
Brief Title: Zinc Supplementation and Nutrition Education Among Children in the Rural Community
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Douala (Other)
Responsible Party: Principal Investigator, NOLLA Nicolas Policarpe, Principal Investigator (Nutrition and Food Science Doctor), University of Douala
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UDouala
Record Dates: First submitted 2020-09-15; First posted 2020-10-05 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Effects of; Serum
MeSH Terms: interventions — Dietary Supplements; Educational Status

STUDY DESIGN:
Intervention Model Description: Evaluation of the anthropometric and biochemistry parameters of children before and after an intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinc supplementation (Experimental): The 25 supplemented children had received an oral dose of 10 mg of zinc sulphate per day for 14 days
  Interventions: Drug: Zinc Supplementation
- Nutrition education of mothers (Experimental): Nutritional information was delivered to each mother to facilitate a change in bad eating habits observed, improve knowledge, attitudes and skills of mothers on child nutrition. The anthropometric and biochemistry parameters of children were taken before and after the maternal nutrition education
  Interventions: Behavioral: Nutrition education of mothers

INTERVENTIONS:
Drug: Zinc Supplementation — The 25 supplemented children had received an oral zinc supplement per day for 14 days and had no dietary restrictions.
  Other Names: Supplementation
  Arms: Zinc supplementation
Behavioral: Nutrition education of mothers — Nutritional information was delivered to each mother to facilitate a change in bad eating habits observed, improve knowledge, attitudes and skills of mothers on child nutrition. The anthropometric and biochemistry parameters of children were taken before and after the maternal nutrition education
  Other Names: Maternal education
  Arms: Nutrition education of mothers

SUMMARY:
Malnutrition among children, especially stunting is a public health problem in Cameroon. This study assesses the impact of zinc supplementation of children and nutrition education of mothers on the nutritional status of the children in the rural community. Dietary surveys, nutritional status, zinc supplementation of children and nutrition education of mothers were carried out. After nutrition education and zinc supplementation, the study showed positive impact of both intervention on the nutritional status of children.

DETAILED DESCRIPTION:
A questionnaire was developed, tested and adjusted prior the field survey. During the study, the knowledge of mothers on child nutrition, the eating habits of children, the estimated consumption of energy, nutrients of children and food availability on the market during harvesting and sowing seasons were evaluated. Moreover, data on zinc supplementation and nutrition education sessions conducted with mothers of these children were collected. The impact of zinc supplementation and maternal education was evaluated by measuring height/age, weight/age and weight/height indices, and levels of serum albumin, calcium, zinc, iron, magnesium and phosphorus before and after interventions.

ELIGIBILITY:
Inclusion Criteria:

* To have an age between 6 to 59 months
* To have signature of informed consent by the parents

Exclusion Criteria:

* To be illnes
* To have severe malnutrition

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2015-12-15 (Actual); Study Completion 2015-12-30 (Actual)

PRIMARY OUTCOMES:
Zinc supplementation among children in the rural community | Zinc supplementation: 14 days
  The supplemented children received the oral zinc sulphate per day for two week and serum zinc concentration were taken before and after the intervention.
Nutrition education of mothers and improvement of nutritionnal status of children | Impact of maternal education: 10 months
  The appropriate information of child nutrition was delivered to each mother. Before and after that maternal nutrition education, the anthropometric and biochemistry parameters of children were mesured.

IPD SHARING:
Plan to Share IPD: No
To share the data with other researchers, we want to publish our study to international review.